CLINICAL TRIAL: NCT05896332
Title: Targeting the Shared Substrates of Alcohol Misuse and Cognitive Impairment: Accelerated rTMS for Older Adults With Alcohol Use Disorder
Brief Title: rTMS in Older Adults With MCI and AUD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00127570; 3P50AA010761-28S1 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder; Mild Cognitive Impairment; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Alcoholism; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: We propose to conduct an open-label Phase I trial of accelerated iTBS-rTMS for AUD+MCI. We propose to recruit 35 treatment-seeking individuals ages 60-85 years, with AUD and cognitive impairment, specifically those meeting criteria for AUD with DSM-5 Mild Neurocognitive Disorder. Individuals will receive 10 sessions of iTBS-rTMS per day, 5 days per week for one week (50 sessions total). All will undergo clinical assessments and brain MRI at pre-treatment and at 1-week post-treatment, and clinical assessments at 4-weeks post-treatment. Weekly post-treatment online self-report assessments will be collected up to four weeks. Resting-state parcellations of pre- and post-fMRI will be completed for personalized targeting and network parcellations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active, Open Label iTBS-rTMS (Experimental): Individuals will receive 10 sessions of iTBS-rTMS per day, 5 days per week for one week (50 sessions total). All will undergo clinical assessments and brain MRI at pre-treatment and at 1-week post-treatment, and clinical assessments at 4-weeks post-treatment. Weekly post-treatment online self-report assessments will be collected up to four weeks. Resting-state parcellations of pre- and post-fMRI will be completed for personalized targeting and network parcellations.
  Interventions: Device: Active, Open Label iTBS-rTMS

INTERVENTIONS:
Device: Active, Open Label iTBS-rTMS — Participants in this group will receive 10 sessions of iTBS-rTMS per day, 5 days per week for one week (50 sessions total)

SUMMARY:
Alcohol misuse is a risk factor for early onset cognitive impairment, contributing to 10% of early onset dementia, with risk corresponding to consumption. Additionally, continued drinking risks worsening cognitive decline and dementia progression, while worsening cognitive impairment contributes to drinking escalation. Repetitive transcranial magnetic stimulation (rTMS) has been shown to improve cognition in Alzheimer's Disease and Related Dimentias (ADRD) and separately reduce heavy drinking in alcohol use disorder. Our objective is to optimize rTMS for simultaneous mitigation of both drinking and cognitive dysfunction in older adults.

DETAILED DESCRIPTION:
Alcohol misuse is a risk factor for early onset cognitive impairment, contributing to 10% of early onset dementia, with risk corresponding to consumption. Additionally, continued drinking risks worsening cognitive decline and dementia progression, while worsening cognitive impairment contributes to drinking escalation. Notably, there exists no intervention targeting the intersection of alcohol misuse and cognitive dysfunction in older adults. It is unclear whether alcohol contributes to a specific form of Alzheimer's Disease and Related Dementias (ADRD) and furthermore whether the impairments and structural brain changes represent classical ADRD neurodegenerative patterns. Despite the unclear etiopathogenesis, there is emerging evidence that repetitive transcranial magnetic stimulation (rTMS) to upregulate executive/cognitive control circuitry can improve cognition in ADRD, and separately reduce heavy drinking in AUD. Our long-term objective is to optimize rTMS for simultaneous mitigation of both drinking and cognitive dysfunction in older adults towards breaking this cycle and thwarting progression to dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85.
* English as a first/primary language.
* Current alcohol use disorder
* Alcohol consumption of at least 4 heavy drinking days (defined as ≥ 4 drinks for women and ≥ 5 for men) per week during the 30-days prior to enrolling;
* Meets actuarial neuropsychological criteria for MCI: ≥2 impaired scores within one cognitive domain, or ≥1 impaired scores in ≥3 domains, where an impaired score is defined as ≤16th percentile using demographically-corrected norms.
* Not pregnant (will administer pregnancy test to confirm)
* Functional visual and auditory acuity to complete all assessments.

Exclusion Criteria:

* Prior diagnosis of Dementia or Major Neurocognitive Disorder per NIA-AA or DSM-5 criteria, and TICS ≤ 22 suggestive of dementia.
* Current substance use disorder other than AUD or nicotine use disorder, bipolar disorder, or schizophrenia spectrum or other psychotic disorder.
* Daily/weekly anticholinergic or sedative use. Stimulants may be allowed pending investigator review. Cholinesterase inhibitors, NMDA receptor antagonists, and antidepressants are allowed if on a stable regimen of 4 weeks prior to enrollment.
* History of significant or unstable condition/s that may impact cognition such as significant cardiac, cerebrovascular, or metabolic disease, developmental disorder, or other neurologic disease (e.g. movement disorder, moderate to severe brain injury, seizures).
* MRI and TMS contraindications (e.g. implants, claustrophobia, conditions/treatments that lower seizure threshold, taking medications that have short half-lives, no identifiable motor threshold).
* Enrolled in a clinical trial or has received an investigational medication or device in the last 30 days.
* Pregnant (will administer pregnancy test to confirm)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in NIH Toolbox-Cognition Battery (NIHTB-CB) Fluid Composite | Week 0 (1 week pre-treatment), Week 2 (immediately post-treatment), Week 6 (4 weeks post-treatment)
  The NIHTB-CB is a performance-based, iPad-administered ~30-minute suite of 7 tests that ascertain abilities in different cognitive domains (i.e. executive function, episodic memory, working memory, processing speed, language). It was developed using advanced psychometric techniques to minimize measurement error and produces normed subtest and composite scores. We will use the fully-corrected T-score (range T=0-100; Mean T=50, SD=10; higher scores indicating better cognition) of the Fluid Cognition Composite (normed for age, sex, years of education, and race/ethnicity) to more accurately reflect global, dynamic thinking abilities that reflect the presence of disease or the impact of interventions, and not premorbid influences on test scores.
Change in Subjective Drinking | Week 0 (1 week pre-treatment), Week 2 (immediately post-treatment), Week 6 (4 weeks post-treatment)
  The Alcohol Timeline Followback (TLFB-90) is a drinking assessment method that obtains estimates of daily drinking. Using a calendar, people provide retrospective estimates of their daily drinking over 90 days from the interview date. Several memory aids can be used to enhance recall (e.g., calendar; key dates serve as anchors for reporting drinking; standard drink conversion).
Change in Network Functional Connectivity between and among cognitive and reward networks and other networks | Week 0 (1 week pre-treatment), Week 2 (immediately post-treatment),
  fMRI will be collected while participants are at rest (i.e. rs-fMRI) during the pre-treatment and post-treatment MRI sessions. The rs-fMRI data will be used to compute functional connectivity, which is the correlation between the activity in each brain region pair over the course of the scan. Each brain region belongs to 1 of 7 previously defined networks (frontoparietal: FPN; default mode: DMN; dorsal attention: DAT; ventral attention: VAT; limbic: LIM; visual: VIS; somatomotor: MOT). Functional connectivity can thus be computed for each network by taking the average of connectivity of all regions belonging to the respective network.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McTeague, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical Univeristy of South Carolina, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05896332/ICF_001.pdf